CLINICAL TRIAL: NCT06650735
Title: Comparison Between Bilateral Lateral Rectus Recession and Bilateral Primary Medial Rectus Resection in Basic Type Intermittent Exotropia
Brief Title: Bilateral Lateral Rectus Recession Versus Bilateral Primary Medial Rectus Resection in Intermittent Exotropia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awadein, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-328-2023
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Intermittent Exotropia
Keywords: IXT; lateral rectus recession; medial rectus resection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMR resection (Active Comparator): Bilateral medial rectus muscle resection
  Interventions: Procedure: BMR resection
- BLR recession (Active Comparator): Bilateral lateral rectus muscle recession
  Interventions: Procedure: BLR recession

INTERVENTIONS:
Procedure: BMR resection — Lid speculum will be applied. Fornix conjunctival incision will be used to expose medial rectus muscle. Area that will be resected will be marked using calipers. Double-armed polyglactin 910 suture (6/0 Vicryl) will be used in securing the muscle.
  The muscle then excised anterior to the sutures and the stump cut flush to the sclera.
  The muscle will be sutured again to the original insertion by scleral sutures which will be tied together.
  Conjunctiva will be closed using polyglactin 910 suture (6/0 Vicryl).
  Arms: BMR resection
Procedure: BLR recession — Lid speculum will be applied. Fornix conjunctival incision will be used to expose lateral rectus muscle. Double-armed polyglactin 910 suture (6/0 Vicryl) will be used in securing the muscle close to the insertion.
  The muscle will then be cut anterior to the sutures flush with the sclera. Calipers will used to mark the new insertion on sclera measured from the stump. The muscle will be sutured again to the new insertion by scleral sutures, which will be tied together.
  Conjunctiva will be closed using polyglactin 910 suture (6/0 Vicryl).
  Arms: BLR recession

SUMMARY:
The goal of this clinical trial is to compare the efficacy of bilateral lateral rectus recession and bilateral primary medial rectus resection in basic type intermittent exotropia

Participants will be randomized into two groups: bilateral lateral rectus (BLR) recession and bilateral medial rectus (BMR) resection groups then followed up in the clinic for 6 months to compare motor alignment and sensory functions

DETAILED DESCRIPTION:
Study location: Cairo university hospitals

Methodology:

Patients with basic type intermittent exotropia who are indicated to undergo surgical intervention will be grouped into two groups one group will undergo bilateral lateral rectus recession and the other will undergo bilateral medial rectus resection.

* Preoperatively, all patients will be subjected to:

  1. A detailed history taking including presence of asthenopia, monocular closure, disfigurement or diplopia. The previous use of glasses for optical correction, use of minus lenses, or prior part time occlusion will be documented.
  2. A detailed ophthalmological examination; including uncorrected and best corrected visual acuity whenever possible, cycloplegic refraction, anterior segment examination and dilated fundus examination.
  3. Motor Evaluation:

     * Ductions and versions will be done to assess the ocular motility in 9 positions of gaze.
     * The angle of deviation will be measured by the alternate prism cover test for both distance (6 meters) and near (33 cm) , with and without glasses.
     * The angles of misalignment will also be measured in side gazes and in straight up and down gaze whenever possible.
     * In patients with near-far disparity, the angle of deviation will be measured again after patching one eye for 30 minutes, as well as after putting +3 D lenses in front of each eye.

     Patients with near-far disparity >10 prism diopters (PD) will not be included
  4. Sensory Evaluation:

     Worth 4 dot test and stereopsis using Random dot test (when possible) The control of exotropia will be assessed using both the newcastle control score

     Patients will be randomly assigned to either surgery using simple randomization by random number generator
* Intervention:

  * One group will undergo bilateral lateral rectus recession and the other will undergo bilateral medial rectus resection according to the standard tables.
  * All cases will be done under general anaesthesia.
  * Both surgeries take about 30 minutes.
  * Postoperative treatment combined tobramycin 0.3% and dexamethasone 0.1% eye drops 3 times daily and the same combination eye ointment at night for 3 weeks.
  * Postoperative follow up will be 1 week, 6 weeks, 3 months and 6 months (minimum follow up)
* Postoperative assessment:

  * Extraocular movement in lateral gazes will be examined for comitance
  * Alignment in the primary position will be assessed and any deviation will be measured using alternate prism cover test
  * Palpebral fissure height will be measured
  * Worth 4 dot test and stereopsis will be assessed (when possible)

    * In cases of failure either over correction or under correction reoperation will be performed after 3 months of the initial surgery.
* Sample size

We are planning a study of the difference in the postoperative angle between the 2 surgical techniques. Assuming a mean difference of 5 PD with a standard deviation of 5 PD, an alpha error of 0.05 and a power of study of 0.8, a total of 17 subjects were found to be needed in each group. Assuming a drop-out rate of 20%, a sample of 20 subjects will be targeted in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with basic type intermittent exotropia
* Measurable angle 25-40 prism diopters

Exclusion Criteria:

* Restrictive or paralytic deviation or if forced duction test is positive on horizontal muscles
* Incomitant deviation, vertical or oblique muscles surgery and significant A or V pattern
* Previous strabismus, orbital or buckle surgery

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Motor alignment in primary position | 12 months
  Success rate defined as orthophoria between exotropia/phoria ≤ to 8 prism diopters & esotropia/phoria ≤ 4 prism diopters

SECONDARY OUTCOMES:
Palpebral fissure height | 12 months
  Change in palpebral fissure height in mm
Lateral gaze comitance/incomitance | 12 months
  Difference between angles of deviation in right gaze, primary position, and left gaze
Stereopsis | 12 months
  Change in stereoacuity in log seconds of arc

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Salah Eldeen Mostafa, MD, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi MY, Hwang JM. The long-term result of slanted medial rectus resection in exotropia of the convergence insufficiency type. Eye (Lond). 2006 Nov;20(11):1279-83. doi: 10.1038/sj.eye.6702095. Epub 2005 Sep 9. PMID 16151478
- [Background] Wang X, Zhang W, Chen B, Liao M, Liu L. Comparison of bilateral medial rectus plication and resection for the treatment of convergence insufficiency-type intermittent exotropia. Acta Ophthalmol. 2019 May;97(3):e448-e453. doi: 10.1111/aos.14056. Epub 2019 Feb 11. PMID 30740923
- [Background] Kushner BJ. Selective surgery for intermittent exotropia based on distance/near differences. Arch Ophthalmol. 1998 Mar;116(3):324-8. doi: 10.1001/archopht.116.3.324. PMID 9514485
- [Background] Pediatric Eye Disease Investigator Group; Writing Committee; Donahue SP, Chandler DL, Holmes JM, Arthur BW, Paysse EA, Wallace DK, Petersen DB, Melia BM, Kraker RT, Miller AM. A Randomized Trial Comparing Bilateral Lateral Rectus Recession versus Unilateral Recess and Resect for Basic-Type Intermittent Exotropia. Ophthalmology. 2019 Feb;126(2):305-317. doi: 10.1016/j.ophtha.2018.08.034. Epub 2018 Sep 3. PMID 30189281